CLINICAL TRIAL: NCT02388555
Title: Coronal Imbalance in Degenerative Lumbar Scoliosis
Brief Title: Perspective Analysis of Coronal Imbalance in Degenerative Scoliosis
Status: Completed | Type: Observational
Sponsor: Nanjing University School of Medicine (Other)
Responsible Party: Principal Investigator, Hongda Bao, Ph.D. candidate, Nanjing University School of Medicine
Other Study IDs: 2013-079-01
Record Dates: First submitted 2015-02-04; First posted 2015-03-17 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Pre-operative group: Respectively recruited patients with DLS. Patients in this group were not surgically treatment. Only pre-operative radiographic parameters were measured.
- Surgically treated group: All DLS patients received posterior osteotomy correction of spinal deformity. The immediate post-operative radiographic measurements were performed.
  Interventions: Procedure: Posterior osteotomy correction

INTERVENTIONS:
Procedure: Posterior osteotomy correction — The DLS patients underwent osteotomy including pedicle subtraction osteotomy (PSO) or Smith-Petersen osteotomy (SPO)
  Groups: Surgically treated group

SUMMARY:
Currently there is paucity of information on the prevalence of pre-operative coronal imbalance in patients with degenerative lumbar scoliosis (DLS) and its influence on surgical outcomes. This study aims to investigate in DLS, the prevalence of coronal imbalance, to propose a novel classification system and to investigate whether pre-operative coronal imbalance affects clinical outcomes following osteotomy. A total of 284 DLS patients were recruited.

DETAILED DESCRIPTION:
A total of 284 DLS patients were recruited into this two-stage study, among which 69 patients were treated by posterior-only correction and the remaining 215 patients received conservative treatment. Using pre-operative long-cassette X-ray films, all patients were classified based on coronal balance distance (CBD) defined as the horizontal distance between C7 plumb line and central sacral vertical line: Type A, CBD < 3cm; Type B, CBD > 3cm and C7PL shifts to the concave side of curve; Type C, CBD > 3cm and C7PL shifts to the convex side of curve. The prevalence of pre-operative coronal imbalance was calculated for stage I study. Post-operative CBD in patients who received surgery was measured to evaluate clinical outcomes for stage II study.

ELIGIBILITY:
Inclusion Criteria:

age > 50 years, diagnosis of DLS based on radiographies and previous medical history and Cobb angle >25°.

Exclusion Criteria:

-

Ages: 50 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with degenerative scoliosis
Sampling Method: Non-Probability Sample
Enrollment: 284 (Actual)
Dates: Start 2010-01; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The relationship between coronal balance classification and immediate post-operative imbalance using radiographic measurements | Up to 3 months
  This part of the study aims to analyze the immediate imbalance after surgery, most of the patients took post-operative films two weeks after surgery, but there were some patients who could not stand at that timepoint and the follow-up time was then at 3 months after surgery.

SECONDARY OUTCOMES:
Relationship between post-operative imbalance and quality of life using quality of life questionnaires including SF-36, ODI and VAS | Up to 1 year
  The quality of life measurements were obtained using questionnaires, and the correlations between coronal imbalance and quality of life were analyzed at 1 year follow-up.
Prevalence of coronal imbalance in degenerative scoliosis using radiographic measurements | Up to 2 year pre-operative follow-up
  The prevalence of coronal imbalance was analyzed in this cross-sectional study. Only a small part of the patients were with longitudinal follow-up. Most of them were without follow-up.